CLINICAL TRIAL: NCT06902454
Title: Evaluation of Crestal Sinus Floor Elevation Using Densah Burs Via Surgical Guide and Simultaneous Implant Placement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa elsbeay, BDS Faculty of Dentistry Tanta University, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tanta U 1712
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: maxillary sinus floor elevation; implant placement; Densah drill

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Densah drill technique for maxillary sinus floor elevation (Experimental): Ten patients with missing maxillary posterior teeth and maxillary sinus pneumatization in this study .the floor of maxillary sinus will be elevated using densah drill via surgical guide with simultaneous implant placement
  Interventions: Device: densah drill technique

INTERVENTIONS:
Device: densah drill technique — ten patients with maxillary sinus pneumatization will be undergo sinus floor elevation using densah drill technique with implant placement

SUMMARY:
Ten patients with missing maxillary posterior teeth and maxillary sinus pneumatization in this study .the floor of maxillary sinus will be elevated using densah drill via surgical guide with simultaneous implant placement . patients will be received, clinically and radiologically examined, and managed at the Oral and Maxillofacial surgery Department, Faculty of Dentistry, Tanta University.

DETAILED DESCRIPTION:
purpose: This study aimed to evaluate maxillary sinus lifting using Densah burs assisted via surgical guide for simultaneous implant installation in atrophic posterior maxilla.

Materials and Methods: Ten patients with missing maxillary posterior teeth and maxillary sinus pneumatization in this study .the floor of maxillary sinus will be elevated using densah drill via surgical guide with simultaneous implant placement The patients will be received, clinically and radiologically examined, and managed at the Oral and Maxillofacial surgery Department, Faculty of Dentistry, Tanta University.

Preoperative evaluation: all patients will be examined clinically and radiographically using Panoramic view to assess the condition of upper and lower jaws mainly bony tissues and Cone beam CT(CBCT) scan to identify the quality and quantity (width, length) of the bone at the surgical site, design and fabricate surgical guide.

Surgical procedure:, a crestal incision will be made and a full thickness mucoperiosteal flap will be elevated, surgical guide will be prepared and adapted to ridge, supported to the neighboring teeth. and the densah drill will be used as the same manner by manufacture ,bone graft will be inserted at the osteotomy site and the implant will be inserted at this site and using osstell ISQ scale to measure implant primary stability. Flap will be sutured using 3-0 vicryl sutures.

Postoperative evaluation: All patients will be followed up at the first week, one month and 4 months postoperatively both clinically if there is pain ,edema , inflamation and radiographically CBCT immediate and 4 months to Detect the amount of elevation will be measured by drawing a tangential line against the implant surface, just above the sinus floor, a measurement will be taken up to the point where the graft material will be seen covering the top of the implant apex ,Detect density of bone graft

ELIGIBILITY:
Inclusion Criteria:

1. Residual bone ridge below the sinus floor ≥ 4 mm ≤6mm.
2. Patients should have no sinus pathology detected radiographically.
3. Inter arch space≥8mm.

Exclusion Criteria:

1. patients with any systemic diseases that affect osseointegration rates.
2. Heavy smokers (>14 cigarettes per day) .
3. pathological lesions in the maxillary sinus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
CBCT for all patients | immediate and after 4 months
  Detect the amount of elevation will be measured by drawing a tangential line against the implant surface, just above the sinus floor, a measurement will be taken up to the point where the graft material will be seen covering the top of the implant apex, Detect density of bone graft

SECONDARY OUTCOMES:
degree of pain evaluated clinically for all patients | one week
  using visual analogue scale:0 represent no pain and 10 represents the highest level of pain
soft tissue healing evaluated clinically for all patients | one week
  presence of dehiscence and exposure of bone or not
infection evaluated clinically for all patients | one week
  presence of signs of infection or not
Evaluation of surgical site for edema | one week
  will be performed using a horizontal and vertical guide with a tape on four reference points: tragus, outer corner of the mouth, outer canthus of the eye and angle of the mandible . The horizontal measure corresponds to the distance between the outer corner of the mouth and the tragus. The vertical measure corresponds to the distance between the outer canthus of the eye and the angle of the mandible. The percentage of facial swelling will be obtained from the difference between measurements made in the immediately and postoperative periods, dividing the result by the value obtained in the immediately period ..

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa El Mostafa, Principal Investigator — faculty of dentistry Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt